CLINICAL TRIAL: NCT05283785
Title: Evaluation of Hand Intrinsic Muscles Functional Recovery After Distal Neurotization of Ulnar Nerve
Brief Title: Ulnar Nerve Neurotization After Ulnar Nerve Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mario Samwel Shawkey Basilios, Resident doctor at orthopedic department , assuit university hospital, Assiut University
Other Study IDs: ulnar nerve neurotization
Record Dates: First submitted 2022-03-02; First posted 2022-03-17 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Ulnar Nerve Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ( group 1): End to End sutures
  Interventions: Procedure: End To End or End to side sutures
- ( group 2 ): End to Side sutures
  Interventions: Procedure: End To End or End to side sutures

INTERVENTIONS:
Procedure: End To End or End to side sutures — End to end or End to side sutures of ulnar nerve by nerve to quadratus muscle ( branch of anterior interosseous nerve )

SUMMARY:
This study will evaluate the hand intrinsic muscles functional recovery after distal neurotization of ulnar nerve

DETAILED DESCRIPTION:
* ulnar nerve injuries result in loss of both the sensory and motor elements within the hand. these injuries can be classified by the site of injury into low injuries and high injuries. In low ulnar nerve injuries, the nerve is injured distal to the motor branch of the Flexor carpi ulnaris (FCU) and motor branch to the Flexor digitorum profundus (FDP) of the ring and little fingers. In low injuries, sensation is lost in palmar ulnar hand and paralysis occurs usually to all 7 interossei, the ulnar 2 lumbrical, the 3 hypothenar, the adductor pollicis, and the deep head of the flexor pollicis brevis muscles .
* After peripheral nerve lesion axonal regeneration is at a rate of 1-2 mm/day. Because muscle fibers undergo irreversible changes after 12 months of denervation, it is important that treatment be undertaken as early as possible for successful functional recovery .
* "Babysitting" nerve fiber transfers can be defined as giving fibers from a healthy donor trunk to a denervated recipient trunk, in order to allow these fibers reach the distal effectors to avoid atrophy; such a procedure has originally been described together with partial neurotomy and has been found to be efficient both in experimental and clinical studies
* As far as it concerns proximal ulnar nerve injuries, babysitting by end-to-side nerve transfer has proven effective in 1 of the 3 series reported, where Colonna et al. analyzed an alternative Martin Grubertype( type of of operation) connection created by a bridge nerve graft between median (donor) and ulnar (recipient) trunks in the distal forearm, which gave interesting, but not ideal results ; "supercharged" reverse end-to side nerve transfers have been reported in latter studies . another person reported 7 cases of distal anterior interosseous to ulnar nerve end-to-end coaptation together with palmar cutaneous branch of the median nerve to the ulnar nerve above the wrist in a previous paper . it has not yet been well-established whether end-to-end or end-to-side gives better results.

nowadays, surgeons performing this type of surgery complain inconsistent outcomes, maybe as an effect of the discrepancy between the number of fibers in donor nerves and those in the recipient one

ELIGIBILITY:
Inclusion Criteria:

1. Site of the injury: at or proximal to level of the elbow
2. Nature of the injury; post traumatic injury.
3. Sex; both males and females.
4. Age; any age.
5. Time of presentation of injury: less than 6 months from injury.

Exclusion Criteria:

1. Any patient with non-post traumatic injury either inflammatory or tumor caused palsy or idiopathic.
2. Any distal injury below origin of FCU branch.
3. Delayed presentation after 6 months of injury.
4. Any patient refusing participation in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. test adductor pollicis muscle.
  2. test palmar inter-osseii.
  3. test dorsal inter-osseii.
  4. test lumbricals.
     * Investigations:
       * Radiological:
         * Plain X-ray
         * EMG and nerve conduction velocity
       * Laboratory : Full laboratory investigations
  Steps of action and techniques used:
  Pre-operative preparation:
  1. recording of pre-existing muscle power,
  2. Clarifying of realistic goals before the surgery,
  3. anti-biotic within 1 hour before surgery> . Surgical techniques transfer of the motor branch of the anterior interosseous nerve that supply pronator quadrates muscle to the motor division of the ulnar nerve ( the deep branch of the ulnar nerve ) by end to end or end to side suture
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
evaluate the hand intrinsic muscles functional recovery after distal neurotization of ulnar nerve | 8 months
  (1) Evaluation of hand intrinsic muscle functional recovery by : A- Muscle power by standard Medical Research Council (MRC) grading B- grip strength by dynamometer C- pinch strength will done based on grading of adductor pollicis muscle. D- Evaluation of clawing will done based on clinical observation E- DASH( Disabilities of the Arm, Shoulder and Hand ) score pre and post

CONTACTS AND LOCATIONS:
Overall Officials: Amr El-Sayed A Ibrahim, Prof Dr, Study Director — Orthopedic and Microsurgery department , assiut university hospital; Yasser M Farouk Ragheb, Lecturar, Study Director — Orthopedic and Microsurgery department , assiut university hospital